CLINICAL TRIAL: NCT04549753
Title: A Study on Brain Activity During Transcranial Direct Current Stimulation for Improving Finger-Hand Function in Stroke Patients
Brief Title: A Study on Brain Activity During Transcranial Direct Current Stimulation in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-04-183
Record Dates: First submitted 2020-09-02; First posted 2020-09-16 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tDCS stimulation group (Experimental): Patients receive four sessions of tDCS stimulation over C3 (patient with left-sided lesion) or C4 (patient with right-sided lesion) based on 10-20 system.
  Interventions: Device: Transcranial direct current simulation

INTERVENTIONS:
Device: Transcranial direct current simulation — Four sessions of stimulation over C3 (patient with left-sided lesion) or C4 (patient with right-sided lesion) based on 10-20 system

SUMMARY:
The purpose of this study is to identify the characteristics of neural plasticity seen in stroke patients by measuring the changes in brain activity during stimulation using functional near-infrared spectroscopy (fNIRS) when applying transcranial direct current stimulation (tDCS) for the purpose of enhancing finger function.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke patients
* Chronic patients over 6 months after onset
* Subcortical stroke
* Patients with the movement of fingers

Exclusion Criteria:

* History of psychiatric disease
* Significant other neurological diseases except for stroke
* Difficult to perform this experiment
* Patients with metal implants
* History of epilepsy
* Pregnancy
* Skin defect at the site of electrode attachment

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in cortical activity using fNIRS signals during brain stimulation | Baseline and about 10 days (immediately after brain stimulation sessions)
  Cortical activities before and after brain stimulation sessions are compared.

SECONDARY OUTCOMES:
Changes in motor evoked potential | Baseline and about 10 days (immediately after brain stimulation sessions)
  Resting motor threshold (rMT) and amplitude of motor evoked potential in first dorsal interosseous muscle are measured. These outcomes are measured by transcranial magnetic stimulation over the motor hotspot. The rMT is defined as the minimum stimulus intensity that produced a minimal motor evoked response at rest. The amplitude means peak to peak of the muscle response.
9-hole pegboard test | Baseline and about 10 days (immediately after brain stimulation sessions)
  The test is a standardized, quantitative assessment used to measure finger dexterity of a patient.
Grip & Tip pinch strength test | Baseline and about 10 days (immediately after brain stimulation sessions)
  The test is to measure the maximum isometric strength of hand, forearm, and finger muscles.
Box & Block test | Baseline and about 10 days (immediately after brain stimulation sessions)
  The test is used to measure the gross manual dexterity of a patient, or of a person using an upper limb prosthetic device.
Fugl-Meyer Assessment | Baseline and about 10 days (immediately after brain stimulation sessions)
  The score is a stroke-specific, performance-based impairment index. The degree of impairment of upper and lower limbs is measured.
Finger tapping test | Baseline and about 10 days (immediately after brain stimulation sessions)
  Response time is measured during finger tapping task.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea